CLINICAL TRIAL: NCT02549690
Title: Effectiveness of Testosterone Gel Pretreatment in Poor Responders Undergoing IVF Treatment: a Randomized Controlled Trial
Brief Title: Testosterone Gel in Poor Responders Undergoing IVF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam National University (Other)
Collaborators: Mỹ Đức Hospital (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Doctor, Vietnam National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCKH/CGRH_ 06_2015
Record Dates: First submitted 2015-09-13; First posted 2015-09-15 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Infertility
Keywords: IVF, Testosterone gel, DHEA, poor responder.
MeSH Terms: conditions — Infertility | interventions — Testosterone; Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone gel (Active Comparator): Testosterone gel 10mg, used transdermally, once a day. Treatment duration: 6-8 weeks
  Interventions: Drug: Testosterone gel
- DHEA (Active Comparator): DHEA 25mg tablet, orally, three times per day. Treatment duration: 6-8 weeks
  Interventions: Drug: DHEA

INTERVENTIONS:
Drug: Testosterone gel — Apply 10mg testosterone gel to the abdomen and rub on with one finger, once a day, in the morning, then allow sites to dry and cover with clothing. Continue the treatment for 6-8 weeks until next IVF treatment.
  Other Names: Androgel
  Arms: Testosterone gel
Drug: DHEA — Take DHEA 25mg tablet orally, three times per day. Continue the treatment for 6-8 weeks, until next IVF treatment.
  Other Names: DHEA tablet
  Arms: DHEA

SUMMARY:
The main purpose of this study is to compare the number of oocytes retrieved after using transdermal testosterone gel 10 mg per day or Dehydroepiandrosterone (DHEA) 75mg per day for 6-8 weeks as pre-treatment for poor ovarian responders undergoing in-vitro fertilization (IVF).

DETAILED DESCRIPTION:
A randomized controlled multiple centers study. The study is designed as a superiority trial. The sample size for this trial of 120 subjects in both groups, based upon the primary endpoint of the number of oocytes retrieved.

IVF patients who have failed to conceive and had poor ovarian response (oocytes retrieved ≤ 3) in the last stimulated cycle though using the maximal dose, which is ≥ 300 IU Follicle-stimulating hormone (FSH) or human menopausal gonadotropin (hMG).

Patients will be randomized to use DHEA or testosterone gel as pretreatment. Randomization will be performed using sealed envelopes developed via a computer generated list with blocks of four. Doctors will be blinded to the randomization, but not patients and nurses.

* Study group 1 use 10 mg transdermal testosterone gel per day.
* Study group 2 use 75mg DHEA per day.

Serum testosterone are measured before treatment. Duration of androgen supplement is 6-8 weeks. After completing the pretreatment, patients are asked to come back when they have menses to begin IVF treatment. Serum testosterone is measured again after the pretreatment in both groups. Patients will be interviewed for side effects and compliance of treatment.

After treatment, patients in both group undergo IVF treatment. IVF treatment will then be performed for all patients, according to the current hospital treatment protocols.

Patients will be followed up until 7th week of gestation, if they have positive pregnancy test after embryo transfer.

Data Analysis and Statistics:

The investigators use Statistical Package for the Social Sciences (SPSS) software 20th version to analyze data. The primary end-point mean of number of retrieved oocytes will be compared between two groups using the Student's t test. The secondary end-points will also be compared between the 2 groups using either the Student's t test or chi-square test.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrolment into this trial, each female subject must fulfill all of the following criteria at the start of enrolment, unless specified otherwise:

* Had one or two previous failure IVF cycle, using GnRH antagonist protocol (≥ 300 IU FSH/hMG per day) and the number of retrieved oocytes are ≤ 3;
* Antral follicle counts (AFC) < 6 or Anti-Mullerian Hormone (AMH) < 1.26 ng/ml

Exclusion Criteria:

To be eligible for enrolment in this study each subject must not meet any of the following criteria:

* Oocyte donation cycle
* Patients have thyroid disease
* Patients have liver or kidney dysfunction
* Patients have abnormal puberty or genital development.
* Patients have previous surgery on ovaries

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes | 30 minutes after oocyte retrieval completed
  Number of oocytes retrieved Number of oocytes retrieved

SECONDARY OUTCOMES:
Clinical pregnancy | 7 weeks after embryo transfer
  Clinical pregnancy is defined by the image gestational sac under ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Linh P Tran, MD, Study Director — Research Center for Genetics and Reproductive Health
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Ward 13. Tan Binh District, Vietnam